CLINICAL TRIAL: NCT05902494
Title: A Retrospective Chart Review of Real-world Treatment Outcomes in Patients With Locally Advanced Unresectable or Metastatic Urothelial Cancer Based on HER2 Expression
Brief Title: HER2 and LA/mUC: A Multi-country Chart Review Cohort Study
Status: Completed | Type: Observational
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Other Study IDs: SGNDV-003; C5731003 (Other: Alias Study Number)
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Cancer; Bladder Cancer; HER2 Mutations; HER2 Overexpression; HER2 Amplification; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to learn about urothelial cancers that make HER2 and how that affects treatment choices for participants with urothelial cancer. During this study, the medical and health records of participants will be reviewed to learn more about their health.

Participants will have urothelial cancer that has grown in the body near where it started (locally advanced) and cannot be removed (unresectable) or has spread through the body (metastatic).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed UC originating from the renal pelvis, ureters, bladder, or urethra. Mixed-cell type tumors are eligible as long as urothelial cell carcinoma is the predominant cell type.
* Locally advanced unresectable or metastatic stage disease
* Formalin fixed paraffin embedded (FFPE) tumor tissue blocks (or freshly sectioned slides, see laboratory manual for details) available for HER2 testing.
* At least 1 prior line of systemic therapy for locally advanced unresectable or metastatic urothelial carcinoma (LA/mUC), including 1 line of platinum-containing chemotherapy.
* Initiation of anticancer therapy for UC after prior progression on platinum-based therapy with or without maintenance avelumab between 01 January 2019 and 12 months before the end of data collection
* Radiographically documented and measurable disease progression immediately before index date

Exclusion Criteria:

* Any concurrent malignant neoplasm requiring systemic therapy during the study window
* Enrollment in a therapeutic clinical trial and received non-standard of care treatment during index line of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults from US and European participating hospitals and physicians' practices with histologically confirmed LA/mUC who initiated therapy after prior progression on platinum-based therapy with or without maintenance avelumab.
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Real-world Objective Response Rate (rwORR) per modified response evaluation criteria in solid tumors version 1.1 (RECIST v1.1) | Up to 5 years
  The proportion of participants who have a best overall response (BOR) based on complete response (CR) or partial response (PR). The BOR for each participant is the best response (radiographically documented and measurable disease or physician-assessed response) achieved after the start date of the lines of treatment (LOT) prior to the initiation of any subsequent LOT.

SECONDARY OUTCOMES:
Percentages of IHC0, 1+, 2+, and 3+ participants | Up to 5 years
Percentages of HER2+ (IHC3+, IHC2+/ISH+), HER2-low (IHC1+, IHC2+/ISH-), HER2-expressing (IHC1+, IHC2+, and IHC3+), and HER2-zero (IHC0) participants | Up to 5 years
Characteristics of LA/mUC participants | Up to 5 years
Real-world Overall Survival (rwOS) | Up to 5 years
  Time from the index date to date of death from any cause.
Characteristics of treatment patterns in LA/mUC participants | Up to 5 years
  Agent, reason for change of LOT, surgery, radiotherapy, number of LOT, treatments in each LOT, mean number of LOT, median time to discontinuation of each LOT
rwORR for each subsequent LOT following the index LOT | Up to 5 years
  The proportion of participants who had a real-world BOR based on CR or PR. The BOR for each participant is the best response (radiographically documented and measurable disease or physician-assessed response) achieved after the start date of the LOT prior to the initiation of any subsequent LOT.
Real-world Time on Treatment (rwTOT) | Up to 5 years
  Time from the start date of the LOT to the end date of the same LOT for any reason.
Real-world Time to Next Treatment (rwTTNT) | Up to 5 years
  The time from the start date of each LOT to the initiation of the next LOT for any reason.
Real-world Progression Free Survival (rwPFS) | Up to 5 years
  Time from the index date to the first recorded disease progression (radiographically documented and measurable disease or physician assessed response) or death from any cause, before the start of next LOT whichever occurs first.
Real-world Duration of Response (rwDOR) | Up to 5 years
  The duration of time from the first documented CR or PR in the LOT to the first recorded disease progression (radiographically documented and measurable disease or physician-assessed response) or death from any cause before the start of the next LOT, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (11):
  - Mayo Clinic, Phoenix, Arizona
  - University of California Irvine, Orange, California
  - Stanford Cancer Institute - School of Medicine, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - University of California Los Angeles, Santa Monica, California
  - University of Colorado Hospital, Aurora, Colorado
  - ICAHN School of Medicine at Mount Sinai,, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Institute - School of Medicine, Durham, North Carolina
  - Avera Cancer Institute Center, Sioux Falls, South Dakota
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
- AKH Wien, Vienna, Austria
- France (8):
  - Chu Bordeaux Hopital Saint Andre, Bordeaux
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Mutualiste Montsouris, Paris
  - CHU LYON, Pierre-Bénite
  - CHU de Rouen., Rouen
  - Foch Hospital, Suresnes
- Germany (3):
  - Alexianer Krefeld GmbH, Krefeld, North Rhine-Westphalia
  - University Hospital Lübeck, Lübeck, Schleswig-Holstein
  - Stuttgart Hospital, Stuttgart

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNDV-003